CLINICAL TRIAL: NCT05407519
Title: A Open-Label, Multi-Center, Single Arm Study to Evaluate the Efficacy and Safety of Tislelizumab Combined With Sitravatinib as Adjuvant Therapy in Participants With Hepatocellular Carcinoma Who Are at High Risk of Recurrence After Curative Hepatic Resection
Brief Title: A Study to Evaluate Tislelizumab Combined With Sitravatinib as Adjuvant Therapy in Participants With HCC at High Risk of Recurrence After Curative Resection
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Collaborators: First Affiliated Hospital Xi'an Jiaotong University (Other); First Affiliated Hospital of Guangxi Medical University (Other); Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, LianxinLiu, Director, Anhui Provincial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-Sitra-2001-IIT
Record Dates: First submitted 2022-05-30; First posted 2022-06-07 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — tislelizumab; sitravatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab 200mg IV q3w + Sitravatinib 100mg PO qd (Experimental): Tislelizumab 200mg IV q3w + Sitravatinib 100mg PO qd Tislelizumab and Sitravatinib will be administered until the disease recurrence, intolerable toxicity, death, withdrawal of consent or completion of 17 cycles of Tislelizumab.
  Interventions: Drug: Tislelizumab + Sitravatinib

INTERVENTIONS:
Drug: Tislelizumab + Sitravatinib — Drug: Tislelizumab Tislelizumab 200mg IV q3w Other Names: BGB-A317, Immunotherapy, Anti-PD-1 antibody Drug: Sitravatinib Sitravatinib 100mg PO qd Other Name: tyrosine kinase inhibitor, TKI

SUMMARY:
This is an open label, multi-center, single arm study to evaluate the efficacy and safety of tislelizumab combined with sitravatinib as adjuvant therapy in hepatocellular carcinoma (HCC) patients who are at high risk of recurrence after curative resection.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is a malignant tumor with high morbidity and mortality. Surgical resection is the most important radical treatment. However, the recurrence rate is high especially in the patients with high risk of recurrence after curative resection. How to reduce postoperative recurrence and improve survival is currently a direction that is worth exploring.

Until now there is no standard postoperative adjuvant therapy. Various adjuvant treatment methods including immunotherapy, targeted therapy, TACE are being studied. This study is to explore the efficacy and safety of tislelizumab combined with sitravatinib as adjuvant therapy in HCC patients who are at high risk of recurrence after curative resection.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with a histopathological or cytologically diagnosis of HCC
2. Subjects who have undergone a curative resection
3. High risk for HCC recurrence as protocol defined
4. No previous systematic treatment and locoregional therapy for HCC
5. Child-Pugh Score, Class A
6. ECOG performance status 0 or 1
7. Full recovery from surgical resection
8. Adequate organ function
9. Absence of major macrovascular invasion
10. No extrahepatic spread
11. Life expectancy of at least 6 months

Exclusion Criteria:

1. Known fibrolamellar HCC, sarcomatoid HCC or mixed cholangiocarcinoma and HCC
2. Evidence of residual, recurrent, or metastatic disease
3. Known history of serious allergy to any component of tislelizumab or sitravatinib preparations
4. History of hepatic encephalopathy
5. Tumor thrombus in portal vein or superior mesenteric vein or inferior caval vein
6. Portal hypertension with bleeding esophageal or gastric varices within 6 months prior to initiation of treatment
7. Any bleeding or thrombotic disorder within 6 months prior to initiation of treatment
8. Any active malignancy within 2 years prior to the start of treatment
9. Active or history of autoimmune disease
10. Other acute or chronic conditions, psychiatric disorders, or laboratory abnormalities that may increase the risk of study participation
11. Pregnant or lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
RFS rate | Observation period 24 months
  2-year Recurrence Free Survival Rate (2-year RFS rate) [Time Frame: Observation period 24 months] 2-year RFS rate is defined as the proportion of patients alive and free of recurrence at 2 years after curative resection.

SECONDARY OUTCOMES:
TTR | 24 months
  1.Time to recurrence (TTR) [Time Frame: 24 months] TTR is defined as the time from the date of curative resection to the first documented recurrence.
RFS | 24 months
  2.Recurrence-Free Survival (RFS) [Time Frame: 24 months] RFS is defined as the time from the date of curative resection to the first documented recurrenceor death due to any cause, whichever occurs first.
RFS rate | 12 months
  3.1-year RFS rate [Time Frame: 12 months]
  1-year RFS rate is defined as the proportion of patients alive and free of recurrence at 1 yearsafter curative resection.
OS | 24 months
  4.Overall Survival (OS）[Time Frame: 24 months] OS is defined as the time from the date of curative resection until death due to any cause.
OS rate | 12 months/24 months
  5.1-year OS rate/2-year OS rate [Time Frame: 12 months/24 months] OS rate is defined as the proportion of patients who have not experienced death from any causeat 12 and 24 months after curative resection.
AEs | 24 months
  6.Adverse Events (AEs) [ Time Frame: 24 months ] The grade of AEs and the number of patients with AEs are assessed based on CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Lianxin LIU secretary of the party committee, Principal Investigator — Anhui Provincial Hospital
Locations (1):
- Anhui province hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No